CLINICAL TRIAL: NCT03373656
Title: Study on Compliance, Safety and Effectivity of Vaccination for Children With Hematologic Malignancies or Solid Tumors and Their Parents
Brief Title: Vaccination for Children of H&O and Their Parents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Cancer Group, China (Network)
Collaborators: Shanghai Pudong District Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCGChina-CCSR-V
Record Dates: First submitted 2017-10-18; First posted 2017-12-14 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Vaccination; Hematologic Malignancy; Solid Tumor, Childhood
Keywords: Vaccination; Childhood; Hematologic Malignancy; Solid Tumor; Immune Deficiency
MeSH Terms: conditions — Hematologic Neoplasms; Immunologic Deficiency Syndromes | interventions — Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low antibody titers (Experimental): Antibody titers lower than protection level
  Interventions: Biological: Vaccination
- high antibody titers (Other): Antibody titers higher than protection level
  Interventions: Other: No Vaccination

INTERVENTIONS:
Biological: Vaccination — Patients with higher antibody titers will accept vaccination. There are two vaccines provided in this study:
  hepatitis B vaccine measles-rubella combined vaccine
  Arms: low antibody titers
Other: No Vaccination — Patients with higher antibody titers will NOT accept vaccination. But we will keep monitoring their antibody titers.
  Arms: high antibody titers

SUMMARY:
The purpose of this study is to study on compliance, safety and effectivity of vaccination for children with hematologic malignancies or solid tumors and their parents.

DETAILED DESCRIPTION:
Children with hematologic malignancies or solid tumors are all facing with immune deficiency due to the disease, the chemotherapy, the hematopoietic stem cell transplantation or the splenectomy, which greatly increases their chance to get infectious diseases. In this study, we will assess the compliance of children with hematologic malignancies or solid tumors and their parents to accept vaccination after finishing treatments, follow up with untoward effect questionnaires to assess the safety, obtain the serum of children patients to test antibody titers and assess the effectivity, provide clues for the study of vaccination in children with hematologic malignancies or solid tumors and provide a scientific basis for the formulation and reunification of vaccination programs.

ELIGIBILITY:
Inclusion Criteria:

1. Children patients(≤18 years) who accepted chemotherapy, hematopoietic stem cell transplantation or splenectomy since our study started.
2. No history of hepatitis B and measles, do not suffer from other diseases that affect immune function and allergic diseases.

Exclusion Criteria:

1. Children patients who did not reach clinical remission after treatment, critically ill or eventually died.
2. Patients who used monoclonal antibodies, especially anti-tumor necrosis factors.
3. Intermittent or low-dose chemotherapy or other immunosuppressive drugs users.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of parents of children willing to be vaccinated after receiving relevant knowledge propagation | 2 years
Number of participants with vaccination-related adverse events | 2 years
The level of serum antibody increased after vaccination | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jin Gao, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China